CLINICAL TRIAL: NCT06597071
Title: Use of Oculometric Measures in the Differential Diagnosis of Typical and Atypical Parkinsonian Conditions: a Pilot Study
Brief Title: Parkinson Atypical Rating of Oculometric Patterns Evaluated Routinely
Acronym: PARATROOPER
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraLight (Industry)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL/APD/2024-1
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease; Progressive Supranuclear Palsy(PSP); Multiple System Atrophy
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive; Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parkinson patients (Active Comparator): Patients diagnosed with Parkinson's disease, ages 50-80, Hoehn & Yahr scale 1-3
  Interventions: Other: NeuraLight PD
- PSP patients (Active Comparator): Patients diagnosed with PSP, according to actual diagnostic criteria from Höglinger GU et al, 2017.
  Interventions: Other: NeuraLight PSP
- MSA patients (Active Comparator): Patients diagnosed with MSA, according to actual diagnostic criteria from Wenning et al, 2022.
  Interventions: Other: NeuraLight MSA
- Healthy (Active Comparator): Healthy subjects with no neurological diseases or cognition deficits
  Interventions: Other: NeuraLight

INTERVENTIONS:
Other: NeuraLight PD — NeuraLight software-based platform for PD patients
  Arms: Parkinson patients
Other: NeuraLight PSP — NeuraLight software-based platform for PSP patients
  Arms: PSP patients
Other: NeuraLight MSA — NeuraLight software-based platform for MSA patients
  Arms: MSA patients
Other: NeuraLight — NeuraLight software-based platform
  Arms: Healthy

SUMMARY:
This is an observational longitudinal study in 4 cohorts of patients with Parkinsonian syndromes, who are visiting the Movement Disorders outpatient clinics.

The aim of the study is to assess the difference of oculometric measures in different neurodegenerative brain conditions and their accuracy over time, and as compared to clinical diagnosis, in order to find a change over time, difference between subgroups and correlations with accepted clinical endpoints in subjects who meet the inclusion criteria and who provide a signed Informed Consent.

DETAILED DESCRIPTION:
As a part of the study, about 40 subjects will undergo a neurological evaluation including motor and cognitive assessments and a NeuraLight session including oculometric measurements and eye-tracking recordings using a novel software-based platform and an eye-tracking system (Tobii, CE-marked class B approved device). Test duration will be approx. 20 minutes. The oculometric evaluation will occur for at least 50% of the cohort 3 times (at baseline, at 6-months and at 12-month follow-up), and all subjects will be recruited over a period of 9 months. All assessments will be performed during a clinic visit unless authorized to be conducted remotely.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age between 40 and 80 years
* <5 years since disease diagnosis
* Normal or corrected vision
* MOCA score ≥ 20
* Ability to follow instructions
* Willing and able to sign an informed consent form Specific
* PD cohort: Ages 50-80, Hoehn & Yahr scale 1-3
* PSP cohort: diagnosed according to actual diagnostic criteria from Höglinger GU et al, 2017.
* MSA cohort: diagnosed according to actual diagnostic criteria from Wenning et al, 2022.

Exclusion Criteria:

-

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of saccadic latency between subgroups | 12 months
  A difference between saccadic latency among the cohorts, enabling a categorization of different patients in study cohorts (p<0.05)
Change of antisaccadic error rate between subgroups | 12 months
  A difference between antisaccadic error rate (%) among the cohorts, enabling a categorization of different patients in study cohorts (p<0.05)
Change of saccadic latency over time as evaluated during visits | 12 months
  Difference between saccadic latency (ms) as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Change of antisaccadic error rate over time as evaluated during visits | 12 months
  Difference between antisaccadic error rate (%) as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Correlation between MDS-UPDRS score and its parts with saccadic latency | 12 months
  The correlation between the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS, scored 0-to a maximum total of 199, indicating the worst possible disability from PD) and its parts with saccadic latency (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05)
Correlation between UMSARS score and its parts with saccadic latency | 12 months
  The correlation between the Unified Multiple System Atrophy Rating Scale (UMSARS) scored 0-to a maximum total of 48, indicating the worst possible disability from MSA) and its parts with saccadic latency (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05)
Correlation between PSP-CDS and its parts with saccadic latency | 12 months
  The correlation between the Progressive Supranuclear Palsy Clinical Deficits Scale (PSP-CDS) scored 0-to a maximum total of 100, indicating the worst possible disability from MSA) and its parts with saccadic latency (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05)

SECONDARY OUTCOMES:
Correlation between MoCA score and its parts with anti-saccadic error rates | 12 months
  The correlation between the Montreal Cognitive Assessment (MoCA, scored 0- to a total possible score is 30 points, where a score of 26 or above is considered normal) with anti-saccadic error rates (%), measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Montreal Cognitive Assessment (MoCA) at visits
Correlation between MoCA score and its parts with smooth pursuit | 12 months
  The correlation between Montreal Cognitive Assessment (MoCA, scored 0- to a total possible score is 30 points, where a score of 26 or above is considered normal) with smooth pursuit speed (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Montreal Cognitive Assessment (MoCA) at visits

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Mir, MD, Principal Investigator — IBIS (Instituto de Biomedicina de Sevilla), Calle Antonio Maura Montaner, Seville, Spain
Locations (1):
- Instituto de Biomedicina de Sevilla (IBiS), Seville, Spain

REFERENCES:
- [Background] Habibi M, Oertel WH, White BJ, Brien DC, Coe BC, Riek HC, Perkins J, Yep R, Itti L, Timmermann L, Best C, Sittig E, Janzen A, Munoz DP. Eye tracking identifies biomarkers in alpha-synucleinopathies versus progressive supranuclear palsy. J Neurol. 2022 Sep;269(9):4920-4938. doi: 10.1007/s00415-022-11136-5. Epub 2022 Apr 30. PMID 35501501